CLINICAL TRIAL: NCT03659253
Title: HIV Awal (Early) Testing & Treatment Indonesia Project Implementing 'Test and Treat' Strategies for HIV Treatment and Prevention in Key Populations in Indonesia: a Prospective Implementation Research Study (Intervention Phase)
Brief Title: HIV Awal (Early) Testing & Treatment Indonesia Project Intervention Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Udayana University (Other); Hasan Sadikin General Hospital (Other); Yayasan Kertipraja (Unknown); World Health Organization (Other); Sardjito Hospital Yogyakarta (Unknown); Universitas Katholik Atmajaya (Unknown); Universitas Padjadjaran (Other); Kirby Institute (Other Government)
Responsible Party: Principal Investigator, Yanri Wijayanti Subronto, MD, MD,PhD,Sp.PD-KPTI,FINASIM, Gadjah Mada University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: The HATI Project HIV Phase 2
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Oral Fluid Based Self Testing (Experimental): All study participants that received intervention and meet inclusion criteria intervention that will be offered OFT
  Interventions: Diagnostic Test: Oral Fluid Based Self Testing; Procedure: Simplified ART Initiation; Behavioral: SMS REMINDER
- Control Group (No Intervention): All HIV Patients in the clinic that not received any intervention
- Simplified ART Initiation (Experimental): All study participants that received intervention and meet inclusion criteria intervention that will be offered SAI
  Interventions: Procedure: Simplified ART Initiation
- CBO AND BROTHEL-BASED ART SERVICE (Experimental): All patients coming to brothel or Community Based Organization services will be offered to get tested and received ART
  Interventions: Procedure: Simplified ART Initiation; Procedure: CBO AND BROTHEL-BASED ART SERVICE; Behavioral: SMS REMINDER
- SMS Reminder (Experimental): All patients that recently found HIV Positive "HIV Naive" offered to get SMS Reminder
  Interventions: Procedure: Simplified ART Initiation; Behavioral: SMS REMINDER; Procedure: MOTIVATIONAL INTERVIEWING
- Motivational Interviewing (Experimental): PWID in Jakarta and Bandung that recently found HIV Positive or lost to follow up ARV offered MI intervention
  Interventions: Procedure: MOTIVATIONAL INTERVIEWING

INTERVENTIONS:
Diagnostic Test: Oral Fluid Based Self Testing — The intervention will introduce provider supervised and unsupervised self-testing as an option for early HIV diagnosis among MSM community in Denpasar Bali Indonesia.
  Other Names: OFT
  Arms: Oral Fluid Based Self Testing
Procedure: Simplified ART Initiation — In this intervention, there will be a change in the clinical practice of ART initiation. In the current practice, clients are asked to perform full pre-ART laboratory examination (complete blood count, liver and renal function tests) before decision of ART initiation. In this intervention, the study participants who are already confirmed as HIV positive and meet specific clinical criteria (see below) will initiate ART (antiretroviral therapy) immediately (after clients' approval) without having to perform full pre-ART laboratory examination. Here, laboratory criteria for initiating ART will be simplified and specific laboratory examination, I.e. creatinine test will be delayed in two weeks after ART initiation.
  Other Names: SAI
  Arms: CBO AND BROTHEL-BASED ART SERVICE; Oral Fluid Based Self Testing; SMS Reminder; Simplified ART Initiation
Procedure: CBO AND BROTHEL-BASED ART SERVICE — The CBOs involved in this intervention are Kebaya and Vesta. Kebaya is an CBO working for Transgender (TG) community. It serves as community gathering place for TG and others, as HIV testing site on regular bases, and also as shelter for homeless HIV patients. The proposed intervention Is that HATI Project will provide HIV testing and treatment in the community, CBO and brothel in collaboration with nearby Puskesmas.
  Other Names: CBO ART SERVICE
  Arms: CBO AND BROTHEL-BASED ART SERVICE
Behavioral: SMS REMINDER — HATI SMS reminder: short message services as reminders to inform ART patients when to take medication, visit the clinics (1 week before the next visit) and remind if they miss clinic appointment.
  Arms: CBO AND BROTHEL-BASED ART SERVICE; Oral Fluid Based Self Testing; SMS Reminder
Procedure: MOTIVATIONAL INTERVIEWING — The approach used in this intervention is an individual counselling with a MI approach, as it is considered a brief form of therapy have been known to be effective in improving HIV treatment adherence.
  The sessions will be held from 3 to up to 10 MI counselling over 6-month period of intervention. The goal of this intervention is to help PWID gain an understanding of their medication-taking behaviors and the actions necessary to successfully maintain a high level of adherence
  Other Names: MI
  Arms: Motivational Interviewing; SMS Reminder

SUMMARY:
This study will be one of the first to systematically evaluate strategies to improve the implementation of a T&T strategy in a concentrated epidemic in Asia.

HATI Project is an implementation research designed, of which consisted of phase I as observation of available standard practice and data collection and phase II implementation of intervention of intervention designed based on the results of phase I.

The first year observation study showed that there are poor cascade of HIV care. The first is the low coverage of HIV test uptake. Along the HIV test and treatment cascade there are substantial reductions.

Furthermore, In the qualitative analysis we found several reasons for the study population for not coming to the ARV sites after being diagnosed with HIV, e.g. social and administrative reasons such as not possessing ID card and unsuited hospital opening hours, etc. Another important finding was the requested laboratory testing by the physicians prior to ART initiation, such as Levels of Haemoglobin, serum transaminases, creatinine, and chest X-ray (manuscript in preparation).

The aims of the proposed interventions are:

1. Increase uptake of HIV testing
2. Increase uptake of HIV treatment initiation
3. Reduce time from testing to treatment initiation
4. Increase percentage of treatment adherence
5. Reducing loss to follow-up on ART
6. Improve treatment outcomes (virological suppression)

There are five interventions proposed:

1. Oral fluid-based testing (self-testing) as a strategy to overcome barriers of testing
2. Simplification of ART initiation
3. CBOs and Brothel-based ART service
4. SMS reminders to increase treatment adherence
5. Motivational Interviewing Approach to increase treatment uptake & adherence

Study sites of the intervention will be conducted in Denpasar (Bali), Yogyakarta (Special Region of Yogyakarta), Bandung (West Java), and Jakarta

The study population for the intervention phase are the same with the first year observational study, i.e.: Female sex workers (FSW), Gay men and other men who have sex with men (MSM), Waria (or transgender) and People who inject drugs (PWID)

DETAILED DESCRIPTION:
Description of the Each Proposed Interventions After the qualitative research, literature reviews, thorough discussions, and based on practical/ logistic considerations, there are five specific interventions that have been chosen. Each of the intervention will be presented here in the same format, i.e. rationale of the intervention, aims of the intervention, study site and key population, description of the intervention, and evaluation of the intervention.

1. ORAL FLUID BASED TESTING (SELF-TESTING) AS A STRATEGY TO OVERCOME BARRIERS OF TESTING AMONG MSM IN BALI, INDONESIA While in Indonesia facility-based HIV testing and counselling (HTC) has been available widely, studies including the HATI qualitative research found that people still worry about stigma, visibility, and social discrimination. Also some reports mentioned lack of privacy and lengthy waiting time for the result impede people to access facility based testing. Public health effort to increase testing coverage and treatment uptakes is urgently needed. Home based testing kit including oral saliva test for HIV has been available in the international market that could bring more control to the communities in finding out their HIV status. A number of studies have reported that the self-testing strategy is accepted and in many cases preferred, however there is still limited study to evaluate its effectiveness in increasing HTC and treatment uptake.

The aim of intervention : To test whether oral fluid self-testing will increase the uptake HTC in MSM and increase the number of HIV+ve MSM who are aware of their status in Bali, Indonesia Description of intervention The current HIV testing practices in Indonesia is happen in two major settings: VCT clinic settingand Mobile testing; both procedure need the health provider team in minimum consist of a doctor, a nurse, a lab technician/analyst and outreach staffs.

The intervention will be different to above practices as it will add or introduce a new option of HIV diagnosis using oral fluids rapid test that could be conducted by the clients themselves (self-testing).

1. The second year intervention will introduce provider supervised and unsupervised self-testing as an option for early HIV diagnosis among MSM community in Denpasar Bali Indonesia.
2. The intervention will be delivered by outreach workers of Kerti Praja Foundation (YKP) in Denpasar Bali. Currently there are 8 outreach workers for MSM in Denpasar. The main task of the outreach staff would be delivering health communication and education around self-testing procedures, distribute the kits to participants who received the test, supervised the test when participants choose to have supervised test, collect the used kits, conduct follow up counselling procedure of the test results including for participants who choose to have unsupervised or home-based test, and conduct referral of reactive result participants to the VCT clinics for confirmatory test and ART services.
3. Potential subjects will be approached in the outreach setting conducted by outreach workers during a standard outreach works. Every MSM will be offered HTC at VCT clinics or mobile VCT available near to their living or working areas. If the client refuse, outreach worker will offer self-testing option.
4. Steps that will take place if potential subject received the intervention i. Subjects will be given detailed information on how to use the test kit in a standardised information (brochure or video) and counselling session for the use of self-testing kit.

ii. Subjects will be offered a supervised self-testing procedure first and if refused unsupervised self-testing procedure will be offered as second option.

iii. All Reactive Subject during OFT intervention will be referred to Clinic for further confirmatory testing.

Evaluation of the impact of the intervention

1. Primary outcome: The number of MSM tested for HIV during the intervention and the number of MSM testing positive for HIV during the intervention
2. Secondary outcomes:

   1. Proportion of those who refuse regular HTC.
   2. Proportion of taking an HIV self-testing kit (regardless of whether used)
   3. Proportion of reporting a positive HIV self-test result to counsellors
   4. Proportion of confirming the result to VCT clinics
   5. CD4 count at enrolment into HATI before and during intervention (may give an indication if people testing earlier i.e.less late presenters)
3. Data collection:

   As per phase one HATI screening, baseline, ARV and follow-up forms will be completed for all participants enrolled into HATI. An additional flag will be added to identify those who had initially tested positive using self-testing-supervised or unsupervised.
4. Impact of other interventions This intervention will be conducted in Bali in parallel with two other intervention; the 'Simplification of ART initiation' and the 'SMS reminders to increase treatment adherence'. However these two interventions target at people already aware of their HIV status and attending a HATI site for treatment. Whereas oral-self testing will be offered in the outreach setting in MSM unaware of their HIV status. Therefore it should be possible to evaluate this intervention independently of these two other interventions. MSM who subsequently attend a HATI clinic for confirmatory testing and receive a positive results will then be eligible for the other intervention packages.
5. The impact of intervention on the improvement of HIV test coverage in MSM population in Bali will be measured using before and after approach.

   2. SIMPLIFICATION OF ART INITIATION TO INCREASE ART UPTAKE AND REDUCE TIME TO ART INITIATION The observational result at the first year of HATI project in the four sites showed that there is a big number of HIV positive clients did not initiate ART in the corresponding HATI sites. There is also lag time between HIV testing and initiation of ARV treatment among study participants. The first year result also showed difference of this average lag time between different types of test and treatment linkage, i.e. hospital to hospital, puskesmas to hospital, CBO (Vesta) to hospital. This time lag between diagnosed as HIV (or testing HIV positive) and ARV initiation putting risk of transmission to their partner and population. In addition, HATI qualitative study stated that MSM, FSW, and transgender did not really like to be referred. They have limited time to move from one place to another place and it will reduce confidentiality.

A One-stop service (same day, same place) and streamlining ARV initiation either in hospital, puskesmas, or in the NGO and hotspots (brothel) may reduce waiting time to ARV initiation and time of appointments of patients to access HIV treatment in hospital.

One of the main (medical) reasons for "delayed" ART initiation is that clients have to conduct pre-ART laboratory examinations, such as Levels of Haemoglobin, serum transaminases, creatinine, and chest X-ray, of which may be very costly (for those who do not have health insurance scheme) and hamper ART initiation. There is a need to streamline pre-ART laboratory testing.

Based on the low incidence rate of nephrotoxicity due to Tenofovir, the intervention will explore the possibility to initiate ART independent of laboratory tests results and creatinine levels will be tested 2 weeks after ART initiation. If result is normal, patients can continue monthly ART. But if there is an (marked) increased of the creatinine level, we will consider as side effect of Tenofovir, and regiment will be changed accordingly.

The aims of the intervention would be:

1. To increase uptake of ART initiation.
2. To reduce time between testing positive and starting treatment Description of the intervention In this intervention, there will be a change in the clinical practice of ART initiation. In the current practice, clients are asked to perform full pre-ART laboratory examination (complete blood count, liver and renal function tests) before decision of ART initiation. In this intervention, the study participants who are already confirmed as HIV positive and meet specific clinical criteria (see below) will initiate ART (antiretroviral therapy) immediately (after clients' approval) without having to perform full pre-ART laboratory examination. Here, laboratory criteria for initiating ART will be simplified and specific laboratory examination, I.e. creatinine test will be delayed in two weeks after ART initiation.

To attract potential clients, the sites will publicise this intervention to the public. If a client from key population come to HATI hospital and or puskesmas site, they will receive pre-HIV test counselling, HIV test, receive results and immediately initiate ART (if it is HIV positive).

All patients newly found to have HIV, or referred with HIV, will be offered recruitment in HATI, regardless of whether or not they meet the criteria for simplified initiation.

Steps to the intervention are as follow:

1. HIV positive patients will be screened for inclusion criteria and clinical symptoms of Tuberculosis (TB). Those meeting the inclusion criteria and does not have symptoms of TB will immediately given ARV regiment for 14 days. The ART regiment consist of Tenofovir + Lamivudine / Emtricitabine + Efavirens. Tenovofir may occasionally causing renal function disturbance. Patients will be checked for Creatinine level on day 14 (two weeks after ART initiation) to monitor Tenofovir sie-effect. The argument to move the examination of laboratory test (from baseline to two weeks after ART initiation) is that patient will already exposed to the drug (tenovofir) so increased creatinine level may be caused by the Tenofovir.
2. One-two days before their next visit, patient will go for creatinine level laboratory testing
3. On the day of the next visit, patient will present their laboratory finding.

   1. If creatinine level is within normal limit, patient can continue their ARV. They will receive ARV for one month and continue as standard HIV care
   2. If creatinine level is slightly increased, they will be closely observed. They will be advised to drink fluid
   3. If creatinine level is > 1.5 gr/dL, ARV regiment will changed. Patients will be referred to hospital for further evaluation.
4. All patients newly found to have HIV, or referred with HIV, will be offered recruitment in HATI, regardless of whether or not they meet the criteria for simplified initiation
5. All patients will be registered in SIHA HIV test and SIHA ARV

Evaluation of the intervention

1. Primary outcome: The increased number of key population tested for HIV and reduction of time lag between diagnosed with HIV and initiation pf ART.
2. Data collection:

   As per phase one HATI screening, baseline, ARV and follow-up forms will be completed for all participants enrolled into HATI. A flag will be added to the follow-up forms to identify those who qualified for 'Simplification of ARV initiation' and those who did not.
3. Intervention has worked if there is increased number of key population doing HIV testing and there is decreased time between testing and treatment in the second years is shorter than in the first year of this study These intervention outcomes will be compared with result in the first year
4. Impact of other interventions:

This intervention is aimed at increasing the uptake of ARV. The other interventions are addressing different aspects of the HIV cascade (testing and adherence) and therefore should not impact on the main variables used to measure the impact of this intervention.

3. COMMUNITY BASED ORGANIZATION (CBO) AND BROTHEL-BASED ART SERVICE Based on the first year result, there is an urgent need to minimize barrier between HIV testing and ART service sites, one of which is One-Stop Service in CBO and or brothel.

Many HIV NGOs and CBOs in Indonesia already conduct mobile VCT where they facilitate HIV testing in their place or else, in collaboration with a puskesmas. There is, however, no known existing ART initiation conducted at CBO and or brothels, on top of the HIV testing service.

In Yogyakarta, there are two CBOs involved in many HIV programs, i.e. Kebaya and Vesta. Kebaya is an organization for transgenders that collaborate with Puskesmas conducting mobile VCT at its place once a month, whereas Vesta, organisation for men who have sex with men (MSM) conducts mobile VCT every week in collaboration with several Puskesmases depending on schedule availability. Out of the 13 puskesmases, 5 Puskesmas have HIV-trained doctors and provide ART (continuation) in Puskesmas.

The Pasar Kembang (abbreviated as Sarkem) brothel collaborated with a Puskesmas conducting HIV testing every three months and STI testing and treatment every two weeks, held at the multi-function hall of the kampung.

Based on the existing activities in Kebaya, Vesta, and Sarkem brothel, it is thought that it would be feasible and beneficial to develop CBO and brothel as One-stop (same day, same place) HIV diagnosis and ARV treatment site, particularly for key populations.

Aims of the intervention

1. To increase uptake of HIV treatment initiation.
2. To Reduce time between testing positive and starting treatment Description of the intervention In Indonesia, there are numerous numbers of NGO (Non Government Organization) and CBO (Community Based Organization) working on HIV issues but are mostly limited to only providing buddies and or outreach workers. Yet, NGOs and CBOs are very close to the key populations. It is rationale to collaborate with HIV NGO and CBO to provide HIV medical services for key populations in the community. This can be done in the condition that NGO/CBO work together with Puskesmas, and that all medical services are provided by health care personnel of Puskesmas.

The CBOs involved in this intervention are Kebaya and Vesta. Kebaya is an CBO working for Transgender (TG) community. It serves as community gathering place for TG and others, as HIV testing site on regular bases, and also as shelter for homeless HIV patients. For this intervention, Kebaya and Vesta will collaborate with HITI Puskesmas to provide medical service to key populations: MSM, FSW, and Transgenders.

The Pasar Kembang brothel has, for many years, work together with PKBI (Perkumpulan Keluarga Berencana Indonesia / Indonesia Planned Parenthood) providing STI and HIV test in situ. For STI service, it is conducted every two weeks, but HIV testing is only every 1 - 3 months. The proposed intervention Is that HATI Project will provide HIV testing and treatment in the community, CBO and brothel in collaboration with nearby Puskesmas. Several steps and training will be taken before commencing the intervention,

Steps to the intervention in the CBO and Brothel are as follow:

1. Key populations are already informed about the service and are invited to participate.
2. They will go for pre-HIV test counseilng and tested for HIV.
3. All patients newly found to have HIV, or referred with HIV, will be offered recruitment in HATI, regardless of whether or not they meet the criteria for simplified initiation
4. All patients will be registered in SIHA HIV test and SIHA ARV

   Delivery and place of the intervention a. The intervention will be delivered by and in CBO and brothel in collaboration with health care workers from the assigned Puskesmas.

   b. Counseling will be conducted by counselor from Puskesmas and CBO. Analyst, nurse and doctor for HIV testing and ART initiation from Puskesmas.

   c. The intervention will be conducted at Vesta and Kebaya office and at a hall of RW (Balai RW) in brothel area.
   1. Vesta and Kebaya CBOs and Pasar Kembang (Sarkem) brothel.
   2. In CBO office, there were rooms which was provided for every phase of this intervention (e.g. room for HIV testing, Counselling, diagnose/treatment). In the brothel, it will be conducted at Hall of RW's and there were small rooms, which was provided for every phase of this intervention.

      Evaluation of the intervention

   <!-- -->

   1. Primary outcome: The increased number of key population tested for HIV and reduction of time lag between diagnosed with HIV and initiation pf ART.
   2. Data collection:

      As per phase one HATI screening, baseline, ARV and follow-up forms will be completed for all participants enrolled into HATI. A flag will be added to the follow-up forms to identify those who qualified for 'Simplification of ARV initiation' and those who did not.
   3. Intervention has worked if there is increased number of key population doing HIV testing and there is decreased time between testing and treatment in the second years is shorter than in the first year of this study. These intervention outcomes will be compared with result in the first year

   Impact of other interventions:

   This intervention is aimed at increasing the uptake of ARV. The other interventions are addressing different aspects of the HIV cascade (testing and adherence) and therefore should not impact on the main variables used to measure the impact of this intervention.

4. SMS REMINDERS TO INCREASE TREATMENT ADHERENCE ARV treatment failure caused by poor adherence, which also lead to AIDS, development of resistant strains of HIV, and death. HATI qualitative study in 2016 showed that the reasons for non-adherence in patients are occurence of ARV side effects, lack of support from family and service provider, or simply forgetting to take the medication.

Several reviews suggest that behavioral intervention could improve ART adherence even though the effects is rarely durable (Sabine et al, 2015). With substantial growth in the number of mobile phone users, researchers and health practitioners have become increasingly interested in the field of mobile health, or m-health, broadly defined as the use of mobile phone technology to improve the delivery of health services. Usage of short message services (SMS) to promote ART adherence could be a good strategy to maintain patients adherence in Indonesia, since data from World Bank in 2015 showed that there were 132 mobile cellular subscriptions per 100 Indonesian people. From anecdotal observation, majority of HATI patients own mobile phones. HATI project in the intervention phase intends to develop a SMS reminder system that effective to promote good ART adherence in Indonesia setting.

Aims of the intervention : SMS Reminder is aimed to improve patient's adherence.

Description of the intervention

1. All HIV positive client in the study sites are offered to join the SMS reminder intervention.
2. For those who refuse to join SMS intervention will receive standard clinic reminder practice
3. For those who agree to join this intervention will protocol below. HATI SMS reminder: short message services as reminders to inform ART patients when to take medication, visit the clinics (1 week before the next visit) and remind if they miss clinic appointment.

The system will automatically flag when patient visits are due, allow automatic SMS reminders for taking medication and flag patients who miss a visit.

HATI Tracing System:

Tracing for patients whom their SMS status were "not delivered" within a month and who do not come on schedule. The list of patients whom their SMS status were "not delivered" within a month and who missed a visit will be forwarded to the peer support/buddy from CBO previously approved to contact them from the informed consent for them to trace. Tracing management will follow regular practice in every ARV sites.

Evaluation of the intervention

1. Evaluation of the intervention will use 3 relevant indicators from the Early Warning Indicators (EWIs) HIV Drug Resistance from WHO, which have been implemented at almost all hospitals providing ART in Indonesia since 2012.

   1. Indicator 1. On-time pill pickup (EWI 1)
   2. Indicator 2. Retention in care (EWI 2)
   3. Indicator 3. Viral load suppression at 12 months (EWI 3)
2. Outcomes a. Primary outcome: 12 months retention in care b. Viral load suppresion (percentage of viral suppresion within 12 months divided by total study participants) c. Secondary outcome: Self-reported adherence d. Process outcomes: i. Proportion of study participants receive SMS reminders Proportion of study participants requesting to stop receiving SMS reminders ii. Proportion of study participants who come to clinic for on-time pill pick-up iii. self-reported adherence
3. Measurements from current HATI data:

   1. Viral load data in 12 months
   2. Self-reported adherence
   3. Proportion of 12 months retention in care

Impact of other interventions: This intervention is aimed at increasing adherence to ARV. The other interventions are addressing different aspects of the HIV cascade (testing and treatment uptake) and therefore should not impact on the main variables used to measure the impact of this intervention.

5. MOTIVATIONAL INTERVIEWING APPROACH TO INCREASE TREATMENT UPTAKE & ADHERENCE

The first year of HATI project data for PWID in Jakarta shows 72% of PWID who enrolled the study wants to start treatment and only 58% of all PWID enrolling the study still continue the treatment currently. In Bandung, only 55% of PWID who enrolled the study wants to start treatment and only 33% of PWID enrolling the study still continuing treatment. From qualitative data, we see an obvious need for mental health services. People are not initiating treatment for fear of side effects, misguided beliefs on the effects of ART, and fear of stigma and discrimination from immediate family members and the community. Of those that have started treatment and stopped, we saw that they suffered from treatment fatigue/burnout, have some issues related to mental health. For example, especially for the PWID, they often find it difficult to manage drug use and manage ART with different harm reduction programs. These issues are rooted in lack of psychosocial assistance, which need to be addressed.

This particular intervention is designed to improve ART uptake and to increase adherence to ART for PWID, by providing better support for psychosocial issues that may affect ART uptake and adherence. there is no existing study, which showed how this model works in enhancing ART adherence among PWID in Indonesia. Therefore, this study will be the first study to provide a MI intervention and also to train health care provider to deliver the MI for enhancing ARV uptake and adherence.

Aims of the intervention :

MI Intervention aims to increase uptakes of HIV treatment initiation and adherence among PWID using motivational intervention approach Description of the intervention: Motivational Interviewing intervention is a client-centered approach for enhancing motivation to change behaviors or maintain healthy behaviors. In the MI intervention, the providers will guide the clients toward change, but the clients are the center of the intervention, the clients are encouraged and empowered to share their barriers of doing something and therefore to find solutions and make a decision for their situations. In other words, the MI counselors will emphasize the clients' autonomy and freedom in making their decisions. In sum, the aim of MI approach is to raise clients' confidence in voicing their arguments by their self.

The approach used in this intervention is an individual counselling with a MI approach, as it is considered a brief form of therapy have been known to be effective in improving HIV treatment adherence. The sites that will be chosen as intervention sites are Puskesmas Grogol Petamburan and Puskesmas Senin.

The sessions will be held from 3 to up to 10 MI counselling over 6-month period of intervention. The goal of this intervention is to help PWID gain an understanding of their medication-taking behaviors and the actions necessary to successfully maintain a high level of adherence.

Steps of the intervention The MI intervention will be done in four stages as described in the flow chart and narration below Stage 1: Pre-ART Initiation Stage 2: ART Initiation Stage 3: ART adherence maintenance Stage 4: Termination Sessions (in the 6th month of intervention) Evaluation of the intervention We will conduct a baseline and end-line survey or comparison between groups, mainly between first-year/baseline cohort and second-year/intervention cohort. Should this intervention be done initially as a pilot, the comparison group might consist of people not receiving intervention in other HATI sites (non-consent or purposively not provided). We will also plan to conduct a small qualitative study to gather clients and providers' satisfaction and feedback of MI approach by in-depth interviews and focused group discussions. This qualitative study will be conducted and documented separately from this intervention protocol.

In the first year, a thorough evaluation will be done after 6 months of the intervention. The evaluation will use data collected from the previous 6 months, as well as collecting new data to assess the acceptability and appropriateness of the topics in the intervention.

Outcomes of the intervention:

• Primary outcome: Clinical outcome: self-reported ARV adherence, CD4 count, VL result of HATI participants on intervention compared with those not receiving the intervention.

• Secondary outcome: Psychological outcome (Self-efficacy & psychological wellbeing).

Output indicators:

* The number of clients receiving intervention and maintained on treatment in 6 months (retention rate),
* Impact indicators: ARV adherence, lost to follow up, come on time to the ARV appointment, VL and CD4 levels, as well as evaluation of psychological well-being.
* Retention rate of people maintained in the intervention
* Number lost to follow up cases after ARV initiation
* Proportion of cascade stage of intervention

Measurements:

* From current HATI Data: CD 4 count, VL result, 6 month follow up
* Questionnaire to assess self-efficacy and psychological well-being by using DASS.
* Self-reported adherence for PWID using ACTG Adherence Baseline and Follow up Questionnaire

ELIGIBILITY:
Inclusion Criteria:

OFT :

1. Refused HTC testing at clinic or outreach setting?
2. Aged 18 years and over;
3. Not known to be HIV-infected;
4. Self-reported anal sex with a man in the last 12 months;

SAI & CBO

1. WHO clinical stage 1 and 2
2. Age < 50 years old
3. Free of Tuberculosis suspicion (based on TB screening form)
4. Not suffering from uncontrolled hypertension (blood pressure more than 140 mmHg) and or diabetes (clinical history based on patients interview)
5. BMI above 18.5 kg/m2
6. ARV naïve
7. Well informed and agree to receive ARV

SMS Reminder :

1. Age: ≥ 16 years old
2. New HIV positive patients initiating ARV
3. Owning a mobile phone with reliable reception
4. Willing to report to research team whenever changing their phone number during the intervention period.

Motivational Interviewing :

Inclusion criteria for the intervention are:

1. PWID with HIV positive;
2. ARV naïve or have ever received treatment but lost to follow up;
3. HATI participants in first phase (regardless the ARV status) and referred by outreach worker/health care provider for adherence counselling because of low level of ARV adherence
4. 16 years old or older

Exclusion Criteria:

* Known HIV Positive
* Refuse to be included in the intervention

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female Male Transgender
Enrollment: 827 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of virologically suppressed | 12 months
  Proportion of people from each key population who are virologically suppressed 12 months after HIV diagnosis. Analyses will be conducted separately for each key affected population

SECONDARY OUTCOMES:
Quantify and comparing other components of the HIV treatment cascade/continuum of care | 12 months
  To quantify and compare other components of the HIV treatment cascade/continuum of care, including
  * Uptake of HIV testing and retesting
  * Clinical and immunological stage at time of HIV diagnosis
  * Uptake of ART and time to initiation of treatment
  * ART adherence and retention in care
Assess the safety and acceptability of early ART Initiation | 12 months
  To assess the safety and acceptability of early ART initiation, including :
  * ART toxicity
  * Short term incidence of AIDS and mortality in those who do and do not initiate ART
  * Proportion failing on first-line ART by virological criteria
  * Emergence of resistance mutations in those failing first-line ART
  * For those who decline immediate ART, reasons for refusal and barriers to initiation of ART
Assess behavioural aspects of Test and Treat Strategy | 12 months
  To assess behavioural aspects of a T&T strategy, including :
  * Impact of ART initiation on risk behaviour
  * Impact of enhanced community-based intervention package on risk behaviour
Number of participants that virologically suppressed | 12 months
  Total number of virologically suppressed individuals from each key affected population

CONTACTS AND LOCATIONS:
Overall Officials: Yanri W Subronto, PhD, Principal Investigator — Gadjah Mada University
Locations (4):
- Indonesia (4):
  - Yayasan Kerti Praja, Denpasar, Bali
  - Dr. Sardjito Hospital, Yogyakarta Indonesia, Yogyakarta, DI Yogyakarta
  - Atma Jaya HIV-AIDS Research Centre, Jakarta, DKI Jakarta
  - Hasan Sadikin Hospital, Bandung, Indonesia, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No